CLINICAL TRIAL: NCT06374966
Title: Real-world Study of Efficacy and Safety of Zonisamide in add-on Therapy for Patients With Focal Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Children's Hospital (Unknown); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Jinhua Second Hospital (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo Women & Children's Hospital (Other); Yuyao People's Hospital (Other); Huzhou Third People's Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Lishui Country People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0246
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Epilepsies, Partial
Keywords: epilepsy; zonisamide
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Zonisamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with focal epilepsy: who using zonisamide as an add-on anti-seizure drug
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — This is a real-world study，so we prospectively enrolled patients with focal epilepsy suitable for taking zonisamide as an add-on medication

SUMMARY:
Patients were first observed for a 4-week baseline period, which required no medication adjustments and a seizure frequency of greater than or equal to 2 times per 4-week . After the baseline observation period, if the patients met the criteria for enrolment and there were no contraindications, zonisamide was added as an additional therapeutic drug.Clinical data were collected before the initiation of treatment, at 1 month, 3 months and 6 months after taking zonisamide respectively, with regular review of blood tests and urinary ultrasound, and imaging and electrophysiological examinations according to the clinical needs of the patient's actual condition.

DETAILED DESCRIPTION:
1. Before starting zonisamide treatment, a 4-week baseline observation period is required, which needs to meet the following criteria: no medication adjustment and at least 2 times of seizure per 4 weeks.
2. If patients meet the criteria for the baseline period, after the baseline observation period, they are required to complete the blood routine, urine routine, renal function, liver function, ultrasound of the urinary tract, and scale completion (including the QOLIE-31 quality of life scale, GAD-7, C-NDDI-E, Pittsburgh sleep quality, and the Epworth Sleepiness Scale (ESS)) prior to initiating treatment. If the patient still meets the inclusion criteria, zonisamide may be added to the treatment, and the patient's seizures and medications prior to zonisamide treatment will be recorded.
3. Outpatient follow-up and scale filling were carried out in the 1st, 3rd and 6th month of zonisamide treatment, and blood tests were reviewed in the first/third (according to the clinical situation) and sixth month, and urological ultrasound was reviewed in the sixth month, and imaging and electrophysiological examinations were carried out according to the clinical need in the light of the actual situation of the patients, and the changes of seizures and side effects during the medication period were recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the International League Against Epilepsy 2017 diagnostic criteria for epilepsy; and the patient's seizures can be clearly classified as partial seizures according to the seizure classification proposed by the International League Against Epilepsy, including simple partial seizures, complex partial seizures, and secondary generalised seizures;
2. Be greater than or equal to 2 years of age;
3. Have been on antiepileptic medication, and during the 4-week period of the retrospective baseline period, the patient did not medication adjustments and had at least 2 seizures greater than or equal to 2 seizures per 4-week period;
4. The patient demonstrated good compliance and was able to complete the scale assessment and record the epilepsy diary on his/her own or with the assistance of a parent;
5. The informed consent form was signed and dated by the patient or a parent or legal guardian.

Exclusion Criteria:

1. Patients who are allergic to zonisamide ;
2. CT or MRI suggestive of progressive intracranial tumours;
3. Severe mental retardation or severe psychiatric disorders;
4. Patients suffering from serious underlying diseases that can affect brain function, such as heart disease, liver disease, renal disease, haematological disorders, malignant tumours, and patients who are immunocompromised;
5. Ultrasound suggestive of renal stones 6) Pregnant or breastfeeding

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As this is a real-world study,we prospectively enrolled patients with focal epilepsy who are suitable for taking zonisamide as an add-on medication
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effective rate at 6 months of treatment | 6 months
  Effective definition: achievement of clinical seizure freedom or >50% reduction in seizure frequency

SECONDARY OUTCOMES:
Effective rate at 3 months of treatment | 3 months
  Effective definition: achievement of clinical seizure freedom or >50% reduction in seizure frequency
Total time to treatment failure | 6 months
  Total time to treatment failure: number of days from initiation of zonisamide to decision to withdraw zonisamide/add new antiepileptic medication
Incidence of side effects | 6 months
  Record the occurrence of side effects in patients and calculate the probability of each side effect occurring

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Wang, doctorate, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (10):
- China (10):
  - Hangzhou Children's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Third People's Hospital, Huzhou, Zhejiang
  - Jiaxing Second hospital, Jiaxing, Zhejiang
  - Jinhua Second hospital, Jinhua, Zhejiang
  - The Fourth Affilicated Hospital of Zhejiang University School of Medicine, Jinhua, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Ningbo Women And Children's Hospital, Ningbo, Zhejiang
  - Ningbo Medical center Lihuili hospital, Ningbo, Zhejiang
  - Yuyao People's hospital, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: No